CLINICAL TRIAL: NCT06628531
Title: Relationship Between Acute Lung Injury and Pulmonary Hyaluronic Acid Deposition After Subarachnoid Hemorrhage
Brief Title: ALI & Pulmonary HA Deposition After SAH
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xintong Ge, Director, Tianjin Medical University General Hospital
Other Study IDs: IRB2024-YS-425-01
Record Dates: First submitted 2024-09-29; First posted 2024-10-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Subarachnoid Haemorrhage (SAH)
Keywords: Subarachnoid haemorrhage; SAH; acute lung injury; ALI; hyaluronic acid
MeSH Terms: conditions — Subarachnoid Hemorrhage; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchoalveolar lavage fluid and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subarachnoid Hemorrhage (SAH)

SUMMARY:
Acute lung injury is a common complication of subarachnoid hematoma (SAH), and a significant risk factor for death in patients with SAH. Unlike neurogenic pulmonary edema and pneumonia following brain injury, the clinical causes of pulmonary injury after SAH are not intracranial hypertension or pulmonary infection. Its occurrence is influenced by the release of catecholamines, the regulatory function of the hypothalamic-pituitary-adrenal (HPA) axis and systemic inflammatory response, but the specific mechanisms are still unclear. Therefore, delving into the pathological mechanisms of SAH-induced lung injury and developing therapeutic strategies based on the findings is of great importance to improve the prognosis of patients.

Abnormal accumulation of hyaluronic acid in the lungs has been reported to be closely related to the pathological progression of various pulmonary injury diseases, such as chest trauma, pulmonary infection and chronic obstructive pulmonary disease. From this, the present research is aimed to explore the levels and dynamic changes of hyaluronic acid in the bronchoalveolar lavage fluid and blood of patients with acute lung injury following SAH, and to analyze its correlation with the prognosis of pulmonary complications, thereby providing assistance for the clinical diagnosis and treatment of SAH.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old with independent behavior ability or authorized legal representative.
* A documented diagnosis of SAH within 5 days.
* A Hunt-Hess scale of Ⅳ or Ⅴ.
* Absence of clinical and etiological evidence of pulmonary infection.

Exclusion Criteria:

* Pregnant or lactating women.
* Present history of traumatic brain injury or intracranial hemorrhage.
* Past history of neurological disorders, lung infection within the past six months, cancer, chronic cardiopulmonary diseases, hematological diseases or renal failure.
* Have participated in clinical trials in the past 4 weeks.
* The investigator considers that not appropriate for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Estimated by statistical analysis, a total of 24 subjects were included from patients admitted to the neurosurgical intensive care unit of Tianjin Medical University General Hospital and the intensive care unit of Tianjin Huanhu Hospital due to aneurysmal SAH.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Hyaluronic acid level in bronchoalveolar lavage fluid after SAH | During the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH
  Hyaluronic acid level (ng/ml) in bronchoalveolar lavage fluid at the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH
Inflammatory cytokines levels in bronchoalveolar lavage fluid after SAH | During the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH
  Inflammatory cytokines (IL-1β, TNF-α and IL-10) levels (pg/ml) in bronchoalveolar lavage fluid at the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH

SECONDARY OUTCOMES:
Serum hyaluronic acid level after SAH | During the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH
  Serum hyaluronic acid level (ng/ml) at the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH
Serum inflammatory cytokines levels after SAH | During the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH
  Serum inflammatory cytokines (IL-1β, TNF-α and IL-10) levels (pg/ml) at the acute phase (1-5 days post-onset) and the chronic phase (10-14 days post-onset) of patients with SAH

CONTACTS AND LOCATIONS:
Overall Officials: Xintong Ge, Study Chair — Tianjin Medical University General Hospital; Yadan Li, Principal Investigator — Tianjin Huanhu Hospital; Ye Tian, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT06628531/Prot_SAP_ICF_000.pdf